CLINICAL TRIAL: NCT03410446
Title: A Phase II, Open-label Clinical Trial of Intranasal Ketamine for Depression in Patients With Cancer Receiving Palliative Care (INKeD-PC Study)
Brief Title: Study of Ketamine for Depression in Cancer Patients Receiving Palliative Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INKeD-PC; 16-5754 (Other: UHN REB)
Record Dates: First submitted 2017-12-28; First posted 2018-01-25 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Depression; Cancer; Palliative Care
MeSH Terms: conditions — Depression; Neoplasms | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): Three doses of ketamine will be given intranasal:
  * Dose 1 will be 50 mg on Day 1
  * Dose 2 will be between 50-100 mg on Day 4
  * Dose 3 will be between 50-150 mg on Day 7
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine is a N-methyl-D-aspartate (NMDA) antagonist.

SUMMARY:
This is a phase 2 study of the drug ketamine for the treatment of depression in cancer patients receiving palliative care. The purpose of this study is to see how useful the drug is at decreasing the severity of depression these patients. Ketamine will be given through the nose.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, voluntary informed consent prior to study enrollment. Participants must be capable of consenting to treatment as substitute decision makers will not be allowed to consent to the study on their behalf
* Males and females ≥ 18 years of age
* Patient is receiving palliative care at Princess Margaret Cancer Centre (PM) including all in-patient units and outpatients
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Major Depressive Disorder (MDD), with a current Major Depressive Episode (MDE)
* Depression severity must be in the moderate to severe range, as determined by a Montgomery-Åsberg Depression Rating Scale (MADRS) score greater than or equal to 20
* Participants must have a confirmed diagnosis of cancer and an estimated life expectancy of less than twelve months, as determined by the palliative care physician

Exclusion Criteria:

* Presence of delirium or suspected delirium
* Severe hypertension or severe cardiac decompensation
* Previous stroke history
* History of intolerability, hypersensitivity or allergy to ketamine
* Patients with bipolar disorder, psychotic disorders, substance use disorders or active suicidality based on a Mini-International Neuropsychiatric Interview (MINI) conducted by a delegated physician will also be excluded
* Current symptoms of psychosis or perceptual disturbances of any kind per investigator discretion
* Pregnancy or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Greater than 25% of participants achieving a clinical response | Day 8
  Montgomery-Åsberg Depression Rating Scale (MADRS) score decreasing by >50%

CONTACTS AND LOCATIONS:
Overall Officials: Madeline Li, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada